CLINICAL TRIAL: NCT05818787
Title: Effect of Vestibular Perceptual Learning on Vestibular Thresholds and Balance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Dan Merfeld, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R01AG073113 (NIH); 3R01AG073113-02S1 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2023-04-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging
Keywords: Vestibular; Perception; Balance; Falls; Learning

STUDY DESIGN:
Intervention Model Description: Three training paradigms and a placebo control task will be evaluated in 3 cohorts of 10 older adults; each subject will complete the control task and one of the three training tasks. Half of each cohort will begin with the perceptual learning protocol, and half will begin with the placebo; assignment will be randomized. The three training protocols will be: 1) a 0.5 Hz roll tilt training protocol previously shown to reduce roll tilt thresholds, 2) a 0.5 Hz inter-aural (Y-Translation training protocol, and 3) a training protocol that includes half 0.5 Hz roll tilts and half 0.5 Hz inter-aural translation.
Who Masked: Outcomes Assessor
Masking Description: Statistical analysis at the conclusion of the trial will be completed using de-identified data, masking the outcomes assessor from the identity and group assignment of each individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Training Protocol 1 - Roll-Tilt Intervention First (Experimental): Participants will complete a roll tilt training protocol previously shown to reduce roll tilt thresholds. The training stimulus parameters are as follows: stimulus size for 0.5 Hz roll tilt motion will be adjusted based upon subject responses using a 2-down, 1-up (2D/1U) staircase, and both auditory and visual feedback will be provided.The training protocol will be completed first, followed by the placebo intervention.
  Interventions: Behavioral: Roll Tilt Training; Behavioral: Placebo Control
- Training Protocol 1 - Placebo First (Experimental): Participants will complete a roll tilt training protocol previously shown to reduce roll tilt thresholds. The training stimulus parameters are as follows: 0.5 Hz roll tilt motion, stimulus size will be adjusted based upon subject responses using a 2D/1U staircase, and both auditory and visual feedback will be provided. The placebo intervention will be completed first, followed by the roll tilt training intervention.
  Interventions: Behavioral: Roll Tilt Training; Behavioral: Placebo Control
- Training Protocol 2 - Y-Translation Intervention First (Experimental): Participants will complete an inter-aural translation training protocol. The training stimulus parameters are as follows: 0.5 Hz inter-aural translation motion, stimulus size will be adjusted based upon subject responses using a 2-down, 1-up (2D/1U) staircase, and both auditory and visual feedback will be provided.The training protocol will be completed first, followed by the placebo intervention.
  Interventions: Behavioral: Translation Training; Behavioral: Placebo Control
- Training Protocol 2 - Placebo First (Experimental): Participants will complete an inter-aural training protocol. The training stimulus parameters are as follows: 0.5 Hz inter-aural translation motion, stimulus size will be adjusted based upon subject responses using a 2D/1U staircase, and auditory and visual feedback will be provided. The placebo intervention will be completed first, followed by the training intervention.
  Interventions: Behavioral: Translation Training; Behavioral: Placebo Control
- Training Protocol 3 - Mixed Intervention First (Experimental): Participants will complete a training protocol that includes half roll tilt and half inter-aural translation. The training stimulus parameters are as follows: 0.5 Hz inter-aural translation motion and 0.5Hz roll tilt, stimulus size will be adjusted based upon subject responses using 2-down, 1-up (2D/1U) staircases, and both auditory and visual feedback will be provided. The training protocol will be completed first, followed by the placebo intervention.
  Interventions: Behavioral: Both Tilt and Translation Training; Behavioral: Placebo Control
- Training Protocol 3 - Placebo First (Experimental): Participants will complete a training protocol that includes half roll tilt and half inter-aural translation. The training stimulus parameters are as follows: 0.5 Hz inter-aural translation motion and 0.5 Hz roll tilt, stimulus size will be adjusted based upon subject responses using 2D/1U staircases, and auditory and visual feedback will be provided. The placebo intervention will be completed first, followed by the training intervention.
  Interventions: Behavioral: Both Tilt and Translation Training; Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Roll Tilt Training — The participants will be tilted and asked to indicate their perceived direction of self-motion (e.g., left or right). Feedback will be provided to promote learning (i.e., improved perception of motion). Feedback will only be provided after the subject response, and thus vestibular (i.e., self-motion) perception is required to judge the direction of the tilt stimulus. After each trial, a three second period of rest will be given. Each day of training will include four blocks of one-hundred trials each. Testing will take place in the dark (except for aims where a visual cue is provided). Subjects will be seated on a motion platform with a 5-point harness and the head restrained. Insert earbuds (along with a white noise signal) will be used to reduce external noise. Subjects will always be asked to make a decision (e.g. left versus right) by pressing buttons with their left or right hands. If not certain, subjects are instructed to provide their best guess.
  Arms: Training Protocol 1 - Placebo First; Training Protocol 1 - Roll-Tilt Intervention First
Behavioral: Translation Training — The participants will be translated and asked to indicate their perceived direction of self-motion (e.g., left or right). Feedback will be provided to promote learning (i.e., improved perception of motion). Feedback will only be provided after the subject responds, and thus vestibular (i.e., self-motion) perception is required to judge the direction of the translation stimulus. After each trial, a three second period of rest will be given. Each day of training will include four blocks of one hundred trials each. Testing will take place in the dark (except for aims where a visual cue is provided). Subjects will be seated on a motion platform with a 5-point harness and the head restrained. Insert earbuds (along with a white noise signal) will be used to reduce external noise. Subjects will always be asked to make a decision (e.g. left versus right) by pressing buttons with their left or right hands. If not certain, subjects are instructed to provide their best guess.
  Arms: Training Protocol 2 - Placebo First; Training Protocol 2 - Y-Translation Intervention First
Behavioral: Both Tilt and Translation Training — The participants will be equally tilted and translated and asked to indicate their perceived direction of self-motion (e.g., left or right) . Feedback will be provided to promote learning (i.e., improved perception of motion). Feedback will only be provided after the subject responds. After each trial, a three second period of rest will be given. Each day of training will include four blocks; 2 blocks of roll tilt and 2 blocks of translation - one hundred trials each. Testing will take place in the dark (except for aims where a visual cue is provided). Subjects will be seated on a motion platform with a 5-point harness and the head restrained. Insert earbuds (along with a white noise signal) will be used to reduce external noise. Subjects will always be asked to make a decision (e.g. left versus right) by pressing buttons with their left or right hands. If not certain, subjects are instructed to provide their best guess.
  Arms: Training Protocol 3 - Mixed Intervention First; Training Protocol 3 - Placebo First
Behavioral: Placebo Control — Participants will complete home-based exercises that are not associated with improving vestibular perception or balance (e.g. saccades, smooth pursuit). Participants will sit in a comfortable chair facing out into a living space. They will then find a stationary object to the right and to the left of themselves as well as above and below their line of sight. Without moving their heads, they will look back and forth and up and down between the objects. Participants will complete a total of 400 eye motions per day for six days.

SUMMARY:
The intervention being studied is a minimal risk perceptual learning protocol delivered in an academic laboratory setting; the goal of the intervention is to improve the perception of passive whole-body tilts and/or translations, as well as balance, by providing feedback following passive tilts or translations of the body. The protocol lasts a total of ~45 days: Day 1 includes a pre-test assessment of perception and balance, as well as 100 repetitions of training, Days 2-7 each include 400 repetitions of training, and Day 6 includes only post-test assessments of perception and balance.

DETAILED DESCRIPTION:
Three training paradigms will be evaluated in 3 cohorts of older 10 adults (N=30; Ages 65 to 89). Motion for all three training paradigms will be provided by a 12" Moog 6DoF motion platform. The first training protocol will be a roll tilt training protocol previously shown to reduce roll tilt thresholds. The second training protocols will be an inter-aural translation training protocol. The third training protocol will include half roll tilt training and half inter-aural translation training. As such, each cohort will perform perceptual training using a combination of the following training parameters:

1. Tilt Training: Training stimuli will be either a roll tilt to the left or right.
2. Translation Training: Training stimuli will be either a translation to the left or right.
3. Both Tilt Training and Translation Training will include half roll tilt training and half inter-aural translation training.
4. Older adults will train using a (A) 2-Down/1-Up (i.e., the size of the tilt stimulus decreases after 2 consecutive correct responses and increases after each incorrect response),
5. Feedback Method: During training, the accuracy of perceptual judgement (e.g., recognizing a left vs. right tilt motion) will be provided to the subject using a combination of auditory feedback and visual feedback. Auditory feedback will inform the subject whether they were correct or incorrect; visual feedback will be provided by the return motion with eyes open and lights on.

The targeted dates for each assessment and intervention period are shown, however, to permit greater adherence to the study protocol, tests of retention will be accepted if they occur within 7 to 10 days after the post-test (for the one-week follow-up) or 30 to 40 days after the post-test (for the one-month follow-up).

1. Intervention-First arm:

   1. Day 1: Pre-test assessment
   2. Days 2-7: Active perceptual learning intervention
   3. Day 8: Post-test assessment
   4. Day 15: One-week retention assessment
   5. Day 38: One-month retention assessment
   6. Days 39-44: Control intervention
   7. Day 45: Post-test assessment
2. Control-First arm:

   1. Day 1: Pre-test assessment
   2. Days 2-7: Control intervention
   3. Day 8: Post-test / Pre-Test assessment
   4. Days 9 to 14: Active perceptual learning intervention
   5. Day 15: Post-test assessment
   6. Day 22: One-week retention assessment
   7. Day 45: One-month retention assessment

ELIGIBILITY:
Inclusion Criteria:

* Must be able to stand
* No leg or foot amputations
* No lower limb braces
* Not currently feeling dizzy/lightheaded
* Not currently pregnant by self-report
* Weight <= 275 pounds

Exclusion Criteria:

* Severe head trauma or traumatic brain injury
* Any vestibular disorder (e.g., Meniere's Disease, Vestibular Migraine, Unresolved benign paroxysmal positional vertigo (BPPV), Vestibular hypofunction, except that due to aging, PPPD) as assessed by a Vestibular OtoNeurologist and Neurotologist using clinical diagnostic tests described in proposal plus any additional clinical evaluations they identify
* History of seizures
* Neurologic illness or condition determined by an Otoneurologist known to impact vestibular or balance function(e.g., stroke, neurodegenerative disorders, demyelinating illness)
* Major psychiatric (e.g., panic disorder, psychosis, etc.) disorder
* Any of the following eye diseases or conditions: amblyopia (or "lazy eye") or history of amblyopia, diagnosis of age-related macular degeneration, retina dystrophy, glaucoma, cataracts, or any other eye condition that limits vision to worse than 20/40
* Recent (<6 months) orthopedic injuries of the lower extremities (e.g., plantar fasciitis, ankle, knee or hip injury, back strain/herniated disc, …).
* Upper extremity injuries requiring current sling immobilization
* Recent surgery
* Any other severe health problem (heart disease, pulmonary disease, cancer, etc.).
* Vision in both eyes must be better than 20/40 with best correction
* Due to the potential for nausea with some of the motion stimuli, and to protect fetus and mother, pregnant women will also be excluded from this study
* Since every possible exclusionary factor cannot be predicted, additional exclusion criteria may be required

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Vestibular Roll Tilt Perceptual Thresholds | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Vestibular perceptual thresholds will be measured using forced-choice methodologies; such methods have been used extensively. Passive, whole body tilts will be delivered using a Moog motion platform. Subjects will be tilted in one of two directions (e.g., towards the left or right) in complete darkness and asked to report their perceived direction of motion. All subjects will be seated in a chair with a 5-point harness. The head will be restrained by a standard motorcycle helmet. Insert earbuds will be worn, reducing external noise by about 20 decibels (dB). To mask potential auditory directionality cues, auditory "noise" - uncorrelated with motion (amplitude, direction, or type) - will be applied at 65 dB sound pressure level (SPL). Motion stimuli will consist of single cycles of sinusoidal acceleration using published methods.
Change in Vestibular Translation Perceptual Thresholds | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Vestibular perceptual thresholds will be measured using forced-choice methodologies; such methods have been used extensively. Passive, whole body inter-aural translations will be delivered using a Moog motion platform. Subjects will be translated in one of two directions (e.g., towards the left or right) in complete darkness and asked to report their perceived direction of motion. All subjects will be seated in a chair with a 5-point harness. The head will be restrained by a standard motorcycle helmet. Insert earbuds will be worn, reducing external noise by about 20 decibel (dB); to mask potential auditory directionality cues, auditory "noise" - uncorrelated with motion (amplitude, direction, or type) - will be applied at 65 dB sound pressure level (SPL). Motion stimuli will consist of single cycles of sinusoidal acceleration using published methods.
Change in the Postural Sway During the Modified Romberg Balance Test | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Static stance will be measured using a tri-axial force plate; postural sway will be measured in response to balance challenges including: (1) standing either on a foam or firm surface, (2) with the eyes either open or closed, and (3) with the feet together or in tandem. The center of pressure (COP) root-mean-square-distance will serve as the primary outcome measure describing postural sway.
Change in Postural Sway during the Sensory Organization Test | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  The Sensory Organization Test (SOT) is a standard clinical and research assessment used to quantify quiet stance postural sway in the presence of unreliable visual and proprioceptive feedback. The conditions of the test include (1) eyes open firm surface, 2) eyes closed firm surface, 3) sway referenced vision firm surface, 4) eyes open sway referenced platform, 5) eyes closed sway referenced platform, 6) sway referenced visual surround and platform. Sway-referencing describes a technique used to alter the reliability of proprioceptive and/or visual inputs by tilting the support surface or visual surround to follow the displacement of the CoP. Center of pressure data will be collected in each condition using a tri-axial force plate; each condition will be repeated three times, for 20 seconds each. The root mean square displacement (RMSD) of the CoP will be calculated for each trial, using the median of three trials as the primary outcome.
Change in Postural Sway during Perturbed Balance | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Our perturbed balance test is a research assessment that we have developed to quantify postural sway in response to motion perturbations of the support surface. Vision will always be occluded (e.g., blindfolded). Forces and torques at the support surface will be quantified. Each trial will take about four minutes to complete and will be repeated three times. The root mean square displacement (RMSD) of the center of pressure (CoP) will be calculated for each trial, as will the gain at each perturbation frequency, using the median of three trials as the outcome variable.

SECONDARY OUTCOMES:
Change in the Time to Failure During the Modified Romberg Balance Test | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Static stance will be measured using a tri-axial force plate; postural sway will be measured in response to balance challenges including: (1) standing either on a foam or firm surface, (2) with the eyes either open or closed, and (3) with the feet together or in tandem. If a trial cannot be completed due to a loss of balance, the time at which the loss of balance occurs will be recorded for each condition.
Change in Pass/Fail Performance on the Modified Romberg Balance Test | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Static stance will be measured using a tri-axial force plate; postural sway will be measured in response to balance challenges including: (1) standing either on a foam or firm surface, (2) with the eyes either open or closed, and (3) with the feet together or in tandem. The ability to complete the test (i.e., without a loss of balance) will be recorded.
Change in Gait | Intervention First Group: Days 1, 8, 15, 38, 45; Placebo First Group: Days 1, 8, 15, 22, 45
  Inertial measurement units (IMUs) will be used to collect motion data to quantify spatiotemporal characteristics of gait (i.e. gait velocity, single/double support time, step length, step width, stride length). Participants will wear noise-cancelling headphones that also provide 65 dB SPL of broadband, auditory noise to remove the contributions of environmental auditory feedback. Each participant will walk at a self-selected pace along a straight 117-foot path. They will make an 180° turn at each end and continue to walk for 6 minutes. IMUs will be placed on each ankle, the lumbar spine, neck, and head. The IMUs on the ankles will be used to detect heel-strike and toe-off, so that a custom MATLAB script will quantify the means and variability of each spatiotemporal characteristic of interest. Measurements will include both means and standard deviations of each parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Merfeld, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner AR, Merfeld DM. Influence of Visual Feedback on Roll Tilt Perceptual Training. Otol Neurotol. 2023 Oct 1;44(9):949-955. doi: 10.1097/MAO.0000000000003990. Epub 2023 Aug 15. PMID 37590890
- [Background] Wagner AR, Kobel MJ, Tajino J, Merfeld DM. Improving self-motion perception and balance through roll tilt perceptual training. J Neurophysiol. 2022 Sep 1;128(3):619-633. doi: 10.1152/jn.00092.2022. Epub 2022 Jul 27. PMID 35894439